CLINICAL TRIAL: NCT01238861
Title: A Phase 2b, Dose-ranging Study to Evaluate the Efficacy and Safety of MEDI-563 in Adults With Uncontrolled Asthma
Brief Title: Study to Evaluate the Efficacy and Safety of MEDI-563 in Adults With Uncontrolled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: MedImmune Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP220; 2010-020126-17 (EudraCT Number)
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; Benralizumab; MEDI-563
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Eosinophilic phenotype (EOS+) Placebo (Placebo Comparator): EOS+ (defined as ELEN Index [proprietary mathematical algorithm to predict sputum eosinophil's greater than or equal to 2 percent] positive and/or FeNO [fraction of exhaled nitric oxide] greater than or equal to [>=] 50 parts per billion [ppb]) participants received matching placebo injections subcutaneous injection every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
  Interventions: Other: Placebo
- EOS+ Benralizumab (2 mg) (Experimental): EOS+ participants received single benralizumab 2 milligram (mg) injection subcutaneously every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
  Interventions: Biological: Benralizumab 2 mg
- EOS+ Benralizumab (20 mg) (Experimental): EOS+ participants received single benralizumab 20 mg injection subcutaneously every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
  Interventions: Biological: Benralizumab 20 mg
- EOS+ Benralizumab (100 mg) (Experimental): EOS+ participants received benralizumab 50 mg as two injections subcutaneously every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
  Interventions: Biological: Benralizumab 100 mg
- Non-eosinophil phenotype (EOS-) Placebo (Placebo Comparator): EOS- (defined as ELEN Index negative and FeNO <50 ppb) participants received matching placebo subcutaneous every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
  Interventions: Other: Placebo
- EOS- Benralizumab (100 mg) (Experimental): EOS- participants received benralizumab 50 mg as two injections subcutaneously every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
  Interventions: Biological: Benralizumab 100 mg

INTERVENTIONS:
Biological: Benralizumab 2 mg — EOS+ participants received single benralizumab 2 milligram (mg) injection followed by a single placebo injection subcutaneously.
  Other Names: MEDI-563
  Arms: EOS+ Benralizumab (2 mg)
Biological: Benralizumab 20 mg — EOS+ participants received single benralizumab 20 mg injection followed by a single placebo injection subcutaneously.
  Other Names: MEDI-563
  Arms: EOS+ Benralizumab (20 mg)
Biological: Benralizumab 100 mg — EOS+ and EOS- participants received two benralizumab 50 mg injections subcutaneously.
  Other Names: MEDI-563
  Arms: EOS+ Benralizumab (100 mg); EOS- Benralizumab (100 mg)
Other: Placebo — EOS+ and EOS- participants received two placebo injections subcutaneously.
  Arms: Eosinophilic phenotype (EOS+) Placebo; Non-eosinophil phenotype (EOS-) Placebo

SUMMARY:
The primary objective of the study is to evaluate the effect of multiple-dose subcutaneous administrations of MEDI-563 on adults with uncontrolled asthma.

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the efficacy and safety of multiple-dose (7 doses) subcutaneous administration of benralizumab (MEDI-563) in adult subjects with uncontrolled asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 75 years at the time of screening
* Adequate contraception from screening through end of trial
* Weight of more than (>) 45 kilogram (kg) but less than or equal to (<=) 150 kg (>100 pound [lb] but <=330 lb)
* History of physician-diagnosed asthma for at least 12 months prior to screening
* Physician prescribed daily use of medium-dose or high-dose inhaled corticosteroid(s) (ICS) plus long-acting beta 2 agonist (LABA) for at least 12 months prior to screening
* Willingness to switch to an ICS/LABA combination product
* Dose of other asthma controller medications must be stable for at least 30 days prior to screening
* At least 2 documented asthma exacerbations in the 12 months prior to screening that required use of a systemic corticosteroid burst
* For subjects 65 years of age or older, a chest x-ray (CXR) or chest computed tomography (CT) that is normal for an asthmatic population
* Ability and willingness to complete the study to Week 66, and if needed to Week 92.

Exclusion Criteria:

* Known history of allergy or reaction to any component of the investigational product formulation
* History of anaphylaxis to any biologic therapy
* Unexplained diarrhea within 30 days prior to screening or diagnosis of helminth parasitic infestation within 6 months prior to screening
* Use of immunosuppressive medication within 3 months prior to screening. Chronic oral prednisone or equivalent up to 10 milligram (mg) daily or 20 mg every other day for asthma is allowed
* Oral corticosteroid burst or short-acting systemic corticosteroid within 30 days prior to screening or during the screening/run-in period
* Acute upper or lower respiratory infections requiring antibiotics or antiviral medications within 30 days prior to the screening or during the screening/run-in period
* Receipt of immunoglobulin or blood products within 30 days prior to screening
* Receipt of any marketed or investigational biologic within 4 months or 5 half-lives prior to screening, whichever is longer
* Receipt of any investigational nonbiologic within 30 days or 5 half-lives prior to screening, whichever is longer
* Previously received MEDI-563
* Any clinically relevant abnormal findings in physical examination
* Past history of clinically significant cardiac disease or any electrocardiogram (ECG) abnormality
* Breastfeeding or lactating women
* History of alcohol or drug abuse within 12 months prior to screening
* History of any known primary immunodeficiency disorder
* Positive medical history for hepatitis B or C. Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to enrol
* A positive human immunodeficiency virus (HIV) test or subject taking antiretroviral medications
* History of cigarette smoking more than or equal to (>=) 10 pack-years or smoking within 12 months prior to screening.
* Known exposure to inhaled occupational agents or fumes with an established diagnosis of occupational asthma
* History of cancer, except for basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy >=12 months prior to screening or other malignancies treated with apparent success with curative therapy >=5 years prior to screening
* Stable dose of allergy vaccination regimen for less than 30 days prior to screening
* Subjects unable to demonstrate acceptable inhaler and peak flow meter techniques.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Raible, MD, Study Director — MedImmune LLC
Locations (74):
- United States (27):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Stockton, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Kissimmee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Stockbridge, Georgia
  - Research Site, Normal, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Summit, New Jersey
  - Research Site, Rochester, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Blue Bell, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Boerne, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Seattle, Washington
- Argentina (4):
  - Research Site, Caba
  - Research Site, Ciudad de Buenos Aires
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Brazil (8):
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Juiz de Fora
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Troyan Municipality
- Canada (4):
  - Research Site, Brampton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, La Malbaie, Quebec
  - Research Site, Québec, Quebec
- Research Site, Bogotá, Colombia
- Mexico (6):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, Villahermosa
  - Research Site, Zapopan
- Peru (4):
  - Research Site, Lima
  - Research Site, San Borja
  - Research Site, San Isidro
  - Research Site, Surco
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Ostrów Wielkopolski
  - Research Site, Piła
  - Research Site, Poznan
  - Research Site, Tarnów
  - Research Site, Warsaw
- Russia (7):
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg

REFERENCES:
- [Result] Castro M, Wenzel SE, Bleecker ER, Pizzichini E, Kuna P, Busse WW, Gossage DL, Ward CK, Wu Y, Wang B, Khatry DB, van der Merwe R, Kolbeck R, Molfino NA, Raible DG. Benralizumab, an anti-interleukin 5 receptor alpha monoclonal antibody, versus placebo for uncontrolled eosinophilic asthma: a phase 2b randomised dose-ranging study. Lancet Respir Med. 2014 Nov;2(11):879-890. doi: 10.1016/S2213-2600(14)70201-2. Epub 2014 Oct 8. PMID 25306557
- [Derived] Sridhar S, Liu H, Pham TH, Damera G, Newbold P. Modulation of blood inflammatory markers by benralizumab in patients with eosinophilic airway diseases. Respir Res. 2019 Jan 18;20(1):14. doi: 10.1186/s12931-018-0968-8. PMID 30658649

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were stratified based on the protocol defined eosinophilic phenotype (EOS+ versus EOS-) and inhaled corticosteroid (ICS) use during a 3-week screening period. A total of 964 participants were screened out of which 609 were randomized in the study, and of which 606 participants received at least one dose of investigational product.
Groups:
- Eosinophilic Phenotype (EOS+) Placebo: EOS+ (defined as ELEN Index [proprietary mathematical algorithm to predict sputum eosinophil's greater than or equal to 2 percent] positive and/or FeNO [fraction of exhaled nitric oxide] greater than or equal to [>=] 50 parts per billion [ppb]) participants received matching placebo subcutaneous injection every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
- EOS+ Benralizumab, 2 mg: EOS+ participants received benralizumab 2 milligram (mg) subcutaneous injection every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
- EOS+ Benralizumab, 20 mg: EOS+ participants received benralizumab 20 mg subcutaneous injection every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
- EOS+ Benralizumab, 100 mg: EOS+ participants received benralizumab 50 mg as two subcutaneous injections every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
- Non-eosinophil Phenotype (EOS-) Placebo: EOS- (defined as ELEN Index negative and FeNO <50 ppb) participants received matching placebo subcutaneous injections every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
- EOS- Benralizumab, 100 mg: EOS- participants received benralizumab 50 mg as two subcutaneous injections every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
Period: Overall Study
Arm/Group | Eosinophilic Phenotype (EOS+) Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | EOS+ Benralizumab, 100 mg | Non-eosinophil Phenotype (EOS-) Placebo | EOS- Benralizumab, 100 mg
Started | 80 | 81 | 81 | 82 | 142 | 140
Completed | 69 | 73 | 70 | 69 | 129 | 125
Not Completed | 11 | 8 | 11 | 13 | 13 | 15
Not completed — Lost to Follow-up | 4 | 2 | 3 | 1 | 1 | 2
Not completed — Unplanned surgery | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Did not meet entry ACQ-6 criteria | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Incorrect enrollment/randomization | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Subject traveled to Argentina by 1 year | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Subject moved out of state/area | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Strongyloides stercoralis antibodies + | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Personal problems | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Unable to continue visits | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Serious adverse event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of compliance | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 4 | 8 | 10 | 9

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population included all randomized participants who received any dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eosinophilic Phenotype (EOS+) Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | EOS+ Benralizumab, 100 mg | Non-eosinophil Phenotype (EOS-) Placebo | EOS- Benralizumab, 100 mg | Total
Number analyzed (Participants) | 80 | 81 | 81 | 82 | 142 | 140 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (11.7) | 47.1 (12.8) | 46.6 (13.2) | 47.8 (12.9) | 50.0 (12.3) | 50.0 (11.5) | 48.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 58 | 48 | 60 | 100 | 98 | 417
  Male | 27 | 23 | 33 | 22 | 42 | 42 | 189

OUTCOME MEASURES:

1. Primary Outcome: Annual Asthma Exacerbation Rate (AER) for Eosinophilic Phenotype (EOS+) Participants
Description: The annual asthma exacerbation rate (AER) was calculated as the total number of observed exacerbations in each group up to week 52, divided by total duration of person-year follow-up in each group. An asthma exacerbation is defined as a progressive increase of asthma symptoms (cough, wheeze, chest tightness, and/or shortness of breath) that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 days as prescribed or administered by the investigator or healthcare provider; or 2) participant initiation of systemic corticosteroids (tablets, suspension or injection) for a duration of at least 3 days as outlined in the Asthma Action Plan provided to the participant by the investigator on Day 1.
Time Frame: Week 1 up to Week 52
Population: as for baseline characteristics
Measure: Number; unit: AER events/person-year
Arm/Group | Eosinophilic Phenotype (EOS+) Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | EOS+ Benralizumab, 100 mg
Number analyzed (Participants) | 80 | 81 | 81 | 82
AER events/person-year | 0.57 | 0.65 | 0.37 | 0.34
Statistical Analysis 1: Comparison: Eosinophilic Phenotype (EOS+) Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.781, Poisson Regression Method; Rate Ratio = 1.09, 80% CI 2-sided [0.74 to 1.59] — The p-value was calculated by Poisson regression with over-dispersion adjustment factor. The correction for potential over dispersion was made by Pearson chi-square
Statistical Analysis 2: Comparison: Eosinophilic Phenotype (EOS+) Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.173, Poisson Regression Method; Rate Ratio = 0.64, 80% CI 2-sided [0.42 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Eosinophilic Phenotype (EOS+) Placebo vs EOS+ Benralizumab, 100 mg; Test type: Superiority or Other; p = 0.096, Poisson Regression Method; Rate ratio = 0.59, 80% CI 2-sided [0.40 to 0.89] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Dose Response in EOS+ Participants
Time Frame: Baseline up to Week 66
Population: Due to change in planned analysis after unblinding of study data, dose response was not performed.
Groups:
- EOS+ Placebo: EOS+ participants received two placebo injections subcutaneously.
Arm/Group | EOS+ Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | EOS+ Benralizumab, 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Minimum Observed Serum Trough Concentration for Benralizumab at Steady-State (Ctrough, ss)
Time Frame: Pre-dose (0 hour), Post-dose on Day 1, 6, Week 4, 16, 24, 32, 40, and 52
Population: The Pharmacokinetic (PK) Population included all participants who received at least one dose of benralizumab and had at least one quantifiable PK observation. One participant, randomized to the EOS- placebo group received a single dose of 100 mg benralizumab on Week 16 and was analyzed for PK in the 100 mg benralizumab group.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Groups:
- Benralizumab, 100 mg: EOS+ and EOS- participants received two benralizumab 50 mg injections subcutaneously.
Arm/Group | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab, 100 mg
Number analyzed (Participants) | 81 | 81 | 223
microgram per milliliter | 34.7 (131) | 182 (180) | 869 (665)

4. Secondary Outcome: Dose-Normalized Minimum Observed Serum Trough Concentration for Benralizumab at Steady-State (Ctrough, ssD)
Time Frame: Pre-dose (0 hour), Post-dose on Day 1, 6, Week 4, 16, 24, 32, 40, and 52
Population: The PK Population included all participants who received at least one dose of benralizumab and had at least one quantifiable PK observation. One participant, randomized to the EOS- placebo group received a single dose of 100 mg benralizumab on Week 16 and was analyzed for PK in the 100 mg benralizumab group.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab, 100 mg
Number analyzed (Participants) | 81 | 81 | 223
microgram per milliliter | 17.3 (65.3) | 9.10 (9.02) | 8.69 (6.65)

5. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) to Benralizumab in Eosinophilic Phenotype (EOS+) Participants
Description: Immunogenicity assessment included determination of anti-drug (benralizumab) antibodies in serum samples. ADA positive was defined as a titer >=50 at any point in the study. It was observed at baseline and any visit during the study.
Time Frame: Baseline up to Week 92
Population: The mITT population included all randomized participants who received any dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | EOS+ Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | EOS+ Benralizumab, 100 mg
Number analyzed (Participants) | 80 | 81 | 81 | 82
percentage of participants | 3.8 | 42.0 | 30.9 | 25.6

6. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (6-items) (ACQ-6) Score at Week 52
Description: Asthma Control Questionnaire (ACQ) is a participant-reported questionnaire to assess the asthma control with 6 items assessing night-time waking, symptoms on waking, activity limitation, shortness of breath, wheeze, and rescue short-acting beta agonist use. Each item was rated on a 7-point Likert scale ranging from 0 (no impairment) to 6 (maximum impairment). Overall ACQ score was the mean of the 6 item scores with a score range of 0 (well controlled) to 6 (extremely poor controlled). Data collected on Day 1 prior to dosing was considered as baseline. Results were reported for overall ACQ score. ACQ-6 score was summarized together for all participants.
Time Frame: Baseline up to Week 52
Population: The mITT population included all randomized participants who received any dose of investigational product. Here "n" signifies participants who were evaluable for this measure for the specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EOS- Placebo: EOS- (defined as ELEN Index negative and FeNO <50 ppb) participants received matching placebo subcutaneous injections every 4 weeks for first 3 doses and then every 8 weeks for next 4 doses up to Week 40.
Arm/Group | EOS+ Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | EOS+ Benralizumab, 100 mg | EOS- Placebo | EOS- Benralizumab, 100 mg
Number analyzed (Participants) | 80 | 81 | 81 | 82 | 142 | 140
units on a scale
  Baseline (n=80,80,80,82,142,140) | 2.7479 (0.9762) | 2.6479 (0.9908) | 2.4750 (0.9106) | 2.5346 (0.9728) | 2.4742 (0.8408) | 2.6381 (0.8330)
  Change at Week 52 (n=34,42,40,39,64,73) | -0.8922 (1.1969) | -1.1032 (1.1207) | -1.2500 (1.2247) | -1.1239 (1.2852) | -0.8418 (1.1343) | -1.1295 (1.1301)
Statistical Analysis 1: Comparison: EOS+ Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.125, ANCOVA; P-value was calculated by analysis of covariance (ANCOVA) with treatment, baseline inhaled steroid status and baseline observed value as covariates
Statistical Analysis 2: Comparison: EOS+ Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.074, ANCOVA; P-value was calculated by ANCOVA with treatment, baseline inhaled steroid status and baseline observed value as covariates
Statistical Analysis 3: Comparison: EOS+ Placebo vs EOS+ Benralizumab, 100 mg; Test type: Superiority or Other; p = 0.057, ANCOVA; [statistical method as in outcome 6, analysis 2]
Statistical Analysis 4: Comparison: EOS- Placebo vs EOS- Benralizumab, 100 mg; Test type: Superiority or Other; p = 0.010, ANCOVA; [statistical method as in outcome 6, analysis 2]

7. Secondary Outcome: Change From Baseline in Mean Total Nasal Symptoms Score (TNSS) at Week 52
Description: Total Nasal Symptoms Score (TNSS) is a 3-item questionnaire, the sum of nasal symptoms, namely, nasal obstruction (rhinorrhea), nasal congestion, and nasal itching/sneezing. Each symptom was rated on a scale from 0-3, with 0 representing no symptoms, 1 mild, 2 moderate, and 3 severe symptoms. TNSS score was a summation of the 3 individual nasal symptom. TNSS score could range from 0 to 9 where higher score indicates worsening. Data was summarized by each treatment group. In addition, data was summarized together for "EOS+ and EOS- Placebo" arms and "EOS+ and EOS- benralizumab 100 mg" arms.
Time Frame: Baseline up to Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Benralizumab (100 mg): EOS+ and EOS- participants received two benralizumab 50 mg injections subcutaneously.
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
units on a scale
  Baseline (n=71,27,25,81) | 4.3 (2.0) | 4.8 (2.0) | 5.3 (1.8) | 4.4 (2.1)
  Change at Week 52 (n=89,39,39,106) | -0.4 (2.90) | -0.8 (2.01) | -1.0 (2.96) | -0.8 (2.24)

8. Secondary Outcome: Change From Baseline in Mean Asthma Symptom Diary Score at Week 51-52
Description: Asthma Symptom Diary included 7 questions about the participant symptom and the overall impact of treatment on the disease during the study period. Mean scores of the 7 questions were calculated to identify asthma symptom-free days. Asthma Symptom Diary Scores were analyzed on a bi-weekly basis and compared to baseline scores. Overall symptom score=(daytime frequency score + daytime severity score + nighttime severity score)/3, where total score ranges from 0 to 9. Higher score represents worsening. Mean asthma symptom diary score were summarized together for all participants. Mean asthma symptom diary score were summarized together for all participants. In addition, data was summarized together for "EOS+ and EOS- Placebo" arms and "EOS+ and EOS- benralizumab 100 mg" arms.
Time Frame: Baseline up to Week 51-52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Participants received two placebo injections subcutaneously.
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
units on a scale
  Baseline (n=204,72,74,210) | 1.58 (0.60) | 1.65 (0.65) | 1.60 (0.61) | 1.60 (0.62)
  Change at Week 51-52 (n=111,36,39,111) | -0.37 (0.61) | -0.56 (0.76) | -0.56 (0.69) | -0.53 (0.67)
Statistical Analysis 1: Comparison: Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.131, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = -0.182, 80% CI 2-sided [-0.336 to -0.028]
Statistical Analysis 2: Comparison: Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.126, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = -0.173, 80% CI 2-sided [-0.317 to -0.028]
Statistical Analysis 3: Comparison: Placebo vs Benralizumab (100 mg); Test type: Superiority or Other; p = 0.097, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = -0.140, 80% CI 2-sided [-0.247 to -0.032]

9. Secondary Outcome: Change From Baseline in Rescue Medication Use at Week 51-52
Description: Participants were provided inhalers of the same dose (medium- or high-dose) inhaled corticosteroid (ICS) plus long-acting beta antagonist (LABA) combination product as baseline prophylactic medication and continued with same dose throughout the study. Rescue medications such as short-term beta2 agonists were used as first-line treatment for worsening asthma symptoms. Investigator prescribed additional short term asthma controller medications included additional ICS, theophylline, inhaled cromones or antimuscarinics; if asthma symptoms remained mild but not resolved. If asthma symptoms worsened, participants received an oral corticosteroid burst. All rescue medications use with prophylactic medication (+ prophylactic) and without prophylactic medication (- prophylactic) was recorded in asthma symptom dairy by participant. Rescue medication use was analyzed on a bi-weekly basis and compared to baseline scores.
Time Frame: Baseline up to Week 51-52
Population: The mITT population included all randomized participants who received any dose of investigational product. Here "n" signifies participants who were evaluable for this measure for the specified time point for each arm, respectively. Data was summarized together for "EOS+ and EOS- Placebo" arms and "EOS+ and EOS- benralizumab 100 mg" arms.
Measure: Mean (Standard Deviation); unit: rescue medication per 2 weeks
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
rescue medication per 2 weeks
  Baseline without prophylactic (n=204,72,74,210) | 3.09 (2.55) | 3.57 (3.67) | 3.82 (4.34) | 3.16 (2.82)
  Baseline with prophylactic (n=204,72,74,210) | 4.07 (3.34) | 4.71 (5.56) | 5.24 (6.40) | 4.22 (3.90)
  Change Week 51-52 -prophylactic(n=111,36,39,111) | -1.2540 (2.4571) | -1.4116 (2.8722) | -1.8804 (5.3129) | -1.1589 (2.0086)
  Change Week 51-52 +prophylactic(n=111,36,39,111) | -1.6855 (3.2875) | -1.6810 (4.2247) | -2.5118 (7.6814) | -1.4693 (2.5603)
Statistical Analysis 1: Comparison: Placebo vs EOS+ Benralizumab, 2 mg; Analysis reported for rescue medication use without prophylactic at Week 51-52; Test type: Superiority or Other; p = 0.642, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = -0.174, 80% CI 2-sided [-0.654 to 0.306]
Statistical Analysis 2: Comparison: Placebo vs EOS+ Benralizumab, 20 mg; Analysis reported for rescue medication use without prophylactic at Week 51-52; Test type: Superiority or Other; p = 0.824, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.111, 80% CI 2-sided [-0.533 to 0.756]
Statistical Analysis 3: Comparison: Placebo vs Benralizumab (100 mg); Analysis reported for rescue medication use without prophylactic at Week 51-52; Test type: Superiority or Other; p = 0.910, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.029, 80% CI 2-sided [-0.297 to 0.355]
Statistical Analysis 4: Comparison: Placebo vs EOS+ Benralizumab, 2 mg; Analysis reported for rescue medication use with prophylactic at Week 51-52; Test type: Superiority or Other; p = 0.992, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = -0.004, 80% CI 2-sided [-0.602 to 0.593]
Statistical Analysis 5: Comparison: Placebo vs EOS+ Benralizumab, 20 mg; Analysis reported for rescue medication use with prophylactic at Week 51-52; Test type: Superiority or Other; p = 0.624, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.337, 80% CI 2-sided [-0.548 to 1.222]
Statistical Analysis 6: Comparison: Placebo vs Benralizumab (100 mg); Analysis reported for rescue medication use with prophylactic at Week 51-52; Test type: Superiority or Other; p = 0.645, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.150, 80% CI 2-sided [-0.267 to 0.567]

10. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 52
Description: FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Data was summarized by each treatment group. In addition, data was summarized together for "EOS+ and EOS- Placebo" arms and "EOS+ and EOS- benralizumab 100 mg" arms.
Time Frame: Baseline and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
liters
  Baseline (n=215,80,81,218) | 2.033 (0.669) | 1.978 (0.701) | 2.080 (0.751) | 2.012 (0.672)
  Change at Week 52 (n=150,51,58,160) | 0.0098 (0.3615) | 0.1631 (0.4691) | 0.1847 (0.5234) | 0.0998 (0.3541)
Statistical Analysis 1: Comparison: Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.014, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.157, 80% CI 2-sided [0.076 to 0.237]
Statistical Analysis 2: Comparison: Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.004, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.184, 80% CI 2-sided [0.102 to 0.266]
Statistical Analysis 3: Comparison: Placebo vs Benralizumab (100 mg); Test type: Superiority or Other; p = 0.026, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.091, 80% CI 2-sided [0.039 to 0.143]

11. Secondary Outcome: Change From Baseline in Mean Forced Vital Capacity (FVC) at Week 52
Description: Forced Vital Capacity (FVC) was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | EOS+ Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | EOS+ Benralizumab, 100 mg | EOS- Placebo | EOS- Benralizumab, 100 mg
Number analyzed (Participants) | 80 | 81 | 81 | 82 | 142 | 140
liters
  Baseline (n=80,80,81,82,135,136) | 3.282 (1.030) | 3.069 (0.957) | 3.285 (1.028) | 3.110 (0.851) | 3.043 (0.864) | 3.126 (0.981)
  Change at Week 52 (n=51,51,58,59,99,101) | 0.029 (0.514) | 0.129 (0.565) | 0.190 (0.586) | 0.166 (0.445) | -0.030 (0.426) | 0.056 (0.371)
Statistical Analysis 1: Comparison: EOS+ Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.384, ANCOVA; [statistical method as in outcome 6, analysis 2]
Statistical Analysis 2: Comparison: EOS+ Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.092, ANCOVA; [statistical method as in outcome 6, analysis 2]
Statistical Analysis 3: Comparison: EOS+ Placebo vs EOS+ Benralizumab, 100 mg; Test type: Superiority or Other; p = 0.134, ANCOVA; [statistical method as in outcome 6, analysis 2]
Statistical Analysis 4: Comparison: EOS- Placebo vs EOS- Benralizumab, 100 mg; Test type: Superiority or Other; p = 0.129, ANCOVA; [statistical method as in outcome 6, analysis 2]

12. Secondary Outcome: Change From Baseline in Peak Expiratory Flow (PEF) at Week 52
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. Peak flow testing for PEF was performed while sitting or standing prior to using any medication (if needed) for asthma. Home PEF was determined separately for morning and evening, and were averaged for each participant. Data was summarized by each treatment group. In addition, data was summarized together for "EOS+ and EOS- Placebo" arms and "EOS+ and EOS- benralizumab 100 mg" arms.
Time Frame: Baseline and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
liters per minute
  Baseline (n=215,80,81,218) | 319.3 (104.7) | 325.5 (101.6) | 323.1 (100.8) | 323.8 (101.7)
  Change at Week 52 (n=150,51,58,160) | 13.0 (64.6) | 29.0 (64.1) | 45.9 (95.5) | 26.6 (66.3)

13. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (Standardized Version) (AQLQ[S]) Score at Week 52
Description: AQLQ: a 32-item questionnaire evaluating quality of life of participants with asthma including 4 domains (symptoms, activity limitations, emotional function, and environmental stimuli). Participants were asked to recall their experiences during the previous 2 weeks and to score each of the 32 questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The overall score was calculated as the mean response to all questions. The 4 domain scores were the means of the responses to the questions in each of the domains. Overall AQLQ score and 4 domain scores ranged from 7 (no impairment) to 1 (severe impairment). The AQLQ(S) responses were categorized as improvement (defined as change from baseline >=0.5), no change (defined as change from baseline >= -0.5 to less than [<] 0.5), and worse (defined as change from baseline < -0.5). Data was summarized by each treatment group.
Time Frame: Baseline and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
units on a scale
  Baseline (n=214,78,80,217) | 3.72 (1.04) | 3.72 (1.17) | 3.79 (1.06) | 3.72 (1.01)
  Change at Week 52 (n=88,39,38,105) | 0.9634 (1.3342) | 1.2612 (1.2082) | 1.4474 (1.4262) | 1.1223 (1.2636)
Statistical Analysis 1: Comparison: Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.069, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.404, 80% CI 2-sided [0.121 to 0.687]
Statistical Analysis 2: Comparison: Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.049, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.462, 80% CI 2-sided [0.163 to 0.761]
Statistical Analysis 3: Comparison: Placebo vs Benralizumab (100 mg); Test type: Superiority or Other; p = 0.168, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.238, 80% CI 2-sided [0.017 to 0.459]

14. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions (EQ-5D) Health State Evaluation at Week 52
Description: The utility-based EQ-5D questionnaire comprises of two parts and provides a generic measure of health for clinical and economic appraisal. The health state valuation was the summary score of mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a 3 category scale (no problem, moderate problem, severe problems). Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. Data was summarized by each treatment group. In addition, data was summarized together for "EOS+ and EOS- Placebo" arms and "EOS+ and EOS- benralizumab 100 mg" arms.
Time Frame: Baseline and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
units on a scale
  Baseline (n=213,79,74,209) | 0.7629 (0.2153) | 0.7418 (0.2376) | 0.7877 (0.1878) | 0.7679 (0.1623)
  Change at Week 52 (n=148,58,53,161) | 0.0853 (0.2096) | 0.0822 (0.3137) | 0.1223 (0.2132) | 0.0824 (0.2179)
Statistical Analysis 1: Comparison: Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.510, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = -0.020, 80% CI 2-sided [-0.058 to 0.019]
Statistical Analysis 2: Comparison: Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.113, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.041, 80% CI 2-sided [0.008 to 0.074]
Statistical Analysis 3: Comparison: Placebo vs Benralizumab (100 mg); Test type: Superiority or Other; p = 0.599, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 0.011, 80% CI 2-sided [-0.016 to 0.038]

15. Secondary Outcome: Change From Baseline in EQ-5D Visual Analog Scale (VAS) at Week 52
Description: The utility-based EQ-5D questionnaire comprises of two parts and provides a generic measure of health for clinical and economic appraisal. The EQ-5D VAS was measured from 0 (worst imaginable health state) to 100 (best imaginable health state). Data was summarized by each treatment group. In addition, data was summarized together for "EOS+ and EOS- Placebo" arms and "EOS+ and EOS- benralizumab 100 mg" arms.
Time Frame: Baseline and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
units on a scale
  Baseline (n=213,79,74,208) | 65.0798 (17.8903) | 65.4937 (18.5063) | 64.3378 (18.1427) | 64.6250 (19.7778)
  Change at Week 52 (n=148,58,53,161) | 12.8041 (19.1036) | 12.5517 (20.8008) | 15.4906 (21.7297) | 13.7391 (20.5139)
Statistical Analysis 1: Comparison: Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.871, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = -0.373, 80% CI 2-sided [-3.333 to 2.586]
Statistical Analysis 2: Comparison: Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.227, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 2.857, 80% CI 2-sided [-0.175 to 5.889]
Statistical Analysis 3: Comparison: Placebo vs Benralizumab (100 mg); Test type: Superiority or Other; p = 0.503, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 1.139, 80% CI 2-sided [-1.041 to 3.319]

16. Secondary Outcome: Change From Baseline in Percentage of Nocturnal Awakening-Free Nights at Week 51-52
Description: Percentage of nocturnal awakening-free nights were analyzed on a bi-weekly basis and compared to baseline scores. Data was summarized by each treatment group. In addition, data was summarized together for "EOS+ and EOS- Placebo" arms and "EOS+ and EOS- benralizumab 100 mg" arms.
Time Frame: Baseline up to Week 51-52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent nocturnal awakening-free nights
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
percent nocturnal awakening-free nights
  Baseline (n=204,72,74,210) | 52.05 (36.96) | 45.07 (40.04) | 51.57 (39.72) | 50.92 (37.72)
  Change at Week 51-52 (n=111,36,39,111) | 19.7595 (39.1388) | 27.1749 (41.7342) | 29.6181 (38.4315) | 23.3054 (36.2761)
Statistical Analysis 1: Comparison: Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.550, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 3.907, 80% CI 2-sided [-4.483 to 12.297]
Statistical Analysis 2: Comparison: Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.215, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 7.659, 80% CI 2-sided [-0.262 to 15.579]
Statistical Analysis 3: Comparison: Placebo vs Benralizumab (100 mg); Test type: Superiority or Other; p = 0.413, ANCOVA; [statistical method as in outcome 6, analysis 2]; Mean Difference (Final Values) = 3.540, 80% CI 2-sided [-2.006 to 9.086]

17. Secondary Outcome: Change From Baseline in Mean Fraction Exhaled Nitric Oxide (FeNO) at Week 52
Description: Data was summarized by each treatment group. In addition, data was summarized together for "EOS+ and EOS- Placebo" arms and "EOS+ and EOS- benralizumab 100 mg" arms.
Time Frame: Baseline up to Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Placebo | EOS+ Benralizumab, 2 mg | EOS+ Benralizumab, 20 mg | Benralizumab (100 mg)
Number analyzed (Participants) | 222 | 81 | 81 | 222
parts per billion
  Baseline (n=222,81,81,222) | 26.88 (23.57) | 39.52 (32.67) | 40.79 (31.03) | 26.68 (23.10)
  Change at Week 52 (n=148,57,56,157) | 1.2523 (16.0200) | -3.2222 (33.2543) | -6.1905 (30.1103) | 1.4384 (28.9090)
Statistical Analysis 1: Comparison: Placebo vs EOS+ Benralizumab, 2 mg; Test type: Superiority or Other; p = 0.896, ANCOVA; [statistical method as in outcome 6, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs EOS+ Benralizumab, 20 mg; Test type: Superiority or Other; p = 0.944, ANCOVA; [statistical method as in outcome 6, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Benralizumab (100 mg); Test type: Superiority or Other; p = 0.667, ANCOVA; [statistical method as in outcome 6, analysis 2]

ADVERSE EVENTS:
Time Frame: From initiation of investigational product administration up to Week 92
Description: The safety population included all participants who received any investigational product and had safety data available for analysis. One participant, randomized to the EOS- placebo group received a single dose of 100 mg benralizumab on Week 16 and was analyzed for safety in the 100 mg benralizumab group .
Groups:
- EOS POS Placebo: EOS+ participants received two placebo injections subcutaneously.
- EOS POS Benralizumab 2 mg: EOS+ participants received single benralizumab 2 milligram (mg) injection followed by a single placebo injection subcutaneously.
- EOS POS Benralizumab 20 mg: EOS+ participants received single benralizumab 20 mg injection followed by a single placebo injection subcutaneously.
- EOS POS Benralizumab 100 mg: EOS+ participants received two benralizumab 50 mg injections subcutaneously.
- EOS NEG Placebo: EOS- participants received two placebo injections subcutaneously.
- EOS NEG Benralizumab 100 mg: EOS- participants received two benralizumab 50 mg injections subcutaneously.
Arm/Group | EOS POS Placebo | EOS POS Benralizumab 2 mg | EOS POS Benralizumab 20 mg | EOS POS Benralizumab 100 mg | EOS NEG Placebo | EOS NEG Benralizumab 100 mg
Serious Adverse Events (participants affected / at risk) | 7/80 | 10/81 | 6/81 | 6/82 | 16/141 | 18/141
Other Adverse Events (participants affected / at risk) | 44/80 | 54/81 | 57/81 | 68/82 | 94/141 | 93/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EOS POS Placebo (N=80) | EOS POS Benralizumab 2 mg (N=81) | EOS POS Benralizumab 20 mg (N=81) | EOS POS Benralizumab 100 mg (N=82) | EOS NEG Placebo (N=141) | EOS NEG Benralizumab 100 mg (N=141)
Acute myocardial infarct (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachyca (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4)
Gastrooesophageal reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 3 (3)
Abdominal wound dehiscen (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 8 (14) | 5 (5)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural cellulit (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infe (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung diseas (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Polyarteritis nodosa (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EOS POS Placebo (N=80) | EOS POS Benralizumab 2 mg (N=81) | EOS POS Benralizumab 20 mg (N=81) | EOS POS Benralizumab 100 mg (N=82) | EOS NEG Placebo (N=141) | EOS NEG Benralizumab 100 mg (N=141)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 2 (4) | 8 (17) | 0 (0) | 10 (17)
Influenza (Infections and infestations) | 4 (4) | 3 (5) | 7 (7) | 6 (6) | 10 (11) | 6 (6)
Sinusitis (Infections and infestations) | 3 (6) | 4 (7) | 3 (3) | 2 (3) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Injection site pain (General disorders) | 0 (0) | 6 (6) | 4 (17) | 2 (3) | 6 (12) | 2 (4)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Acute sinusitis (Infections and infestations) | 3 (7) | 4 (6) | 2 (2) | 3 (3) | 2 (4) | 6 (8)
Bronchitis (Infections and infestations) | 3 (4) | 8 (10) | 6 (8) | 3 (4) | 13 (20) | 9 (11)
Nasopharyngitis (Infections and infestations) | 8 (13) | 11 (19) | 7 (13) | 13 (16) | 5 (6) | 13 (17)
Pharyngitis (Infections and infestations) | 3 (3) | 8 (10) | 3 (3) | 7 (9) | 5 (5) | 6 (6)
Rhinitis (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 2 (3) | 5 (5) | 3 (7)
Upper respiratory tract (Infections and infestations) | 4 (6) | 7 (12) | 7 (8) | 5 (6) | 10 (12) | 11 (14)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (3) | 1 (1) | 3 (4) | 5 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 5 (6) | 3 (3) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 2 (2) | 2 (4) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 8 (13) | 8 (13) | 6 (10) | 9 (10) | 8 (9) | 13 (17)
Asthma (Respiratory, thoracic and mediastinal disorders) | 30 (51) | 28 (59) | 24 (42) | 26 (36) | 42 (67) | 42 (77)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (5) | 8 (13) | 6 (8) | 4 (8) | 5 (11)
Hypertension (Vascular disorders) | 1 (2) | 3 (3) | 0 (0) | 3 (3) | 4 (4) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.